CLINICAL TRIAL: NCT07006714
Title: Preoperative Single High-Dose Vitamin D for Correcting Deficiency in Hip and Knee Arthroplasty Patients-A Prospective Study
Brief Title: Preoperative Correction of Vitamin D Deficiency in Total Joint Arthroplasty (TJA)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Michele D'Apuzzo, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20250203
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis; Vitamin D Deficiency
MeSH Terms: conditions — Osteoarthritis; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vitamin D Deficient Group (Experimental): Participants who are vitamin D deficient and undergo standard of care TJA will receive a single dose of vitamin D. Total participation for up to 90 days.
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Patients with a Vitamin D3 level of less than 30 nanograms per milliliter will receive a single oral (pill) dose of 300,000 international units of vitamin D3.

SUMMARY:
The purpose of this study is being conducted to determine whether correcting low levels of vitamin D with a single high-dose supplement reduces complications after the participant's primary TJA.

ELIGIBILITY:
Inclusion Criteria:

* Serum 25(OH)D < 30 ng/mL within 2 weeks of surgery.
* Able to provide informed consent.

Exclusion Criteria:

* Follow-up duration < 90 days anticipated.
* Acute hepatitis, cancer, organ transplant recipients, or dialysis patients.
* Extra vitamin D supplementation within 90 days post-surgery.
* Preoperative serum 25(OH)D ≥ 30 ng/mL.
* Adults unable to consent (excluded).
* Individuals under 18 (excluded).
* Pregnant women (excluded).
* Prisoners (excluded).

Ages: 18 Years to 96 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Prosthetic joint infection as measured by the Musculoskeletal Infection Society (MSIS) criteria. | Up to 90 days.
  The MSIS criteria infection scores range from 0-1 as not infected, 2-5 as possibly infected, and 6 or greater than 6 as infected.

SECONDARY OUTCOMES:
Hospital length of stay | Up to 90 days.
  Measured in hours.
Number of medical complications | Up to 90 days.
  Measured in number.
Number of readmission rates | Up to 90 days.
  Measured in number.

CONTACTS AND LOCATIONS:
Overall Officials: Michele D'Apuzzo, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No